CLINICAL TRIAL: NCT07019090
Title: An Open-label Extension Trial of the Long-term Safety and Efficacy of HSK44459 Tablets in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Long-term Safety and Efficacy Study of HSK44459 Tablets in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: IPF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK44459-204
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK44459 (Experimental)
  Interventions: Drug: HSK44459

INTERVENTIONS:
Drug: HSK44459 — HSK44459

SUMMARY:
This study is open to people with idiopathic pulmonary fibrosis (IPF) . They can only take part if they have completed treatment in a previous study with a medicine called HSK44459.

The primary object of this study is to find out how well people with idiopathic pulmonary fibrosis (IPF) tolerate long- term treatment with HSK44459.

ELIGIBILITY:
Inclusion Criteria:

1.IPF patients who completed the last dose treatment of HSK44459 in previous trials without prematurely discontinuing treatment permanently according to protocol , and have been evaluated by the researchers to have greater benefits than risks, and may benefit from continued treatment with HSK44459

Exclusion Criteria:

1. Patient will plan to undergo lung transplantation.
2. Patients with a Body Mass index (BMI) <18.5 kg/m² that experienced an unexplained and clinically significant (>10%) weight loss during the previous trials.
3. History of malignancy within 5 years prior to screening.
4. History of depression or anxiety disorder.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-27 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events during the study period | Up to 52 weeks

IPD SHARING:
Plan to Share IPD: No